CLINICAL TRIAL: NCT03006471
Title: Effect of Dapagliflozin on Blood Pressure Variability in Patients With Prediabetes and Prehypertension Without Pharmacological Treatment
Brief Title: Effect of Dapagliflozin on Blood Pressure Variability in Prediabetes and Prehypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, PhD, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAPA-BP variability
Record Dates: First submitted 2016-12-13; First posted 2016-12-30 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: PreDiabetes; Prehypertension
Keywords: Prediabetes; Prehypertension; Variability of blood pressure; ABPM; Dapagliflozin; SGLT2
MeSH Terms: conditions — Prediabetic State; Prehypertension | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin capsules, 10 mg, one per day before breakfast during 12 weeks.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo capsules, one per day before breakfast during 12 weeks.
  Interventions: Drug: Placebo - Cap

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg, one per day before breakfast during 12 weeks.
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Placebo - Cap — one per day before breakfast during 12 weeks.
  Other Names: Calcined magnesium
  Arms: Placebo

SUMMARY:
Prediabetes is defined as an intermediate metabolic state that leads to the development of type 2 diabetes mellitus (DM2) and the prehypertension is a category assigned to identify patients who are at risk of developing hypertension (AH), in both pathologies the abnormalities in the variation of blood pressure (BP) has been related to organ damage, its evaluation is performed by ambulatory blood pressure monitoring (ABPM).

Dapagliflozin is a selective and reversible inhibitor of the sodium-glucose co-transporter type 2 (SGLT-2), which reduces renal reabsorption of glucose and promotes the excretion of glucose through the urine, in the way that glucose blood. Another reported effects is the decrease on BP, so it would be interesting to evaluate this effects in patients with prediabetes and prehypertension, as a potential therapy to treat disorders and to prevent progression to DM2 and Hypertension, respectively.

The aim of this study is to evaluate the effect of Dapagliflozin on variability of blood pressure in patients with prediabetes and prehypertension without pharmacological treatment.

The investigators hypothesis is that the administration of dapagliflozin decreases variability of blood pressure in patients with prediabetes and prehypertension without pharmacological treatment.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial in 30 patients with a diagnosis of prediabetes and prehypertension without treatment.

They will be assigned randomly two groups of 15 patients each to receive 10 mg of Dapagliflozin (Forxiga, Astra Zeneca) or placebo, one per day before breakfast during 12 weeks.

There will be calculated body mass index (BMI) and blood pressure variability. This protocol it's already approved by the local ethics committee and written informed consent it's going to be obtained from all volunteers.

Statistical analysis will be presented through measures of central tendency and dispersion, average and deviation standard for quantitative variables; frequencies and percentages for variable qualitative. Qualitative variables will be analyzed by X2/ exact fisher test, will be used for differences inter-group Mann-Whitney U Test and coefficient of variation, Wilcoxon Test and index of variability for the within-groups differences. It will be considered statistical significance p ≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Patients both sexes, age between 30 and 60 years
* Diagnosis of prediabetes according American Diabetes Association criteria (fasting blood glucose levels between 100-126 mg/dl; postprandial blood glucose levels after an oral glucose tolerance test with 75 of oral glucose between 140-199 mg/dl; or glycosylated hemoglobin between 5.7-6.4%)
* Diagnosis of prehypertension according (JNC8) Eighth Joint National Committee blood pressure between 120-139/ 80-89 mmHg.

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Hypersensibility to ingredients of intervention
* Physical impossibility for taking pills
* Known uncontrolled renal, hepatic, heart or thyroid diseased
* Diabetes diagnosis
* Previous treatment for glucose or blood pressure Triglycerides ≥400 mg/dL
* Total cholesterol ≥240 mg/dL
* History of cardiovascular disease
* Worker per shift / night

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL GONZALEZ, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin | Placebo
Started | 15 | 15
Completed | 13 (Two patients did not complete the study due to early withdrawal) | 13 (Two patients did not complete the study due to early withdrawal)
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47 (7) | 50 (5) | 48.5 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 30
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Mexico]
  Mexico | 15 | 15 | 30
Body weight [Mean (Standard Deviation); unit: kg] — The body weight was measured with a bioimpedance balance and the entered values reflect the body weight at baseline
  kg | 74 (10) | 80 (12) | 77 (11)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mas Index was calculated with the Quetelet index formula and the entered values reflect the body mass index at baseline
  kg/m^2 | 30 (2) | 31 (2) | 30.5 (2)
Office Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — The office blood pressure was measured at baseline using the Omron 907-E digital sphygmomanometer (Healthcare, Inc.).
  mmHg | 127 (7) | 127 (5) | 127 (6)
Office Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — The office blood pressure was measured at baseline using the Omron 907-E digital sphygmomanometer (Healthcare, Inc.).
  mmHg | 80.0 (6.0) | 81.0 (7.0) | 80.5 (6.5)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] — The fasting glucose level was evaluated with enzymatic/colorimetric techniques at baseline
  mmol/L | 6.3 (0.3) | 6.0 (0.4) | 6.15 (0.35)
2-hours plasma glucose after a oral glucose tolerance test [Mean (Standard Deviation); unit: mmol/L] — 2-hours glucose was evaluated with an oral glucose tolerance test (75 g of glucose load) using enzymatic/colorimetric technique at baseline
  mmol/L | 8.4 (1.4) | 7.9 (2.4) | 8.15 (1.9)
Glycated hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: percentage of A1C] — Glycosylated hemoglobin was evaluated at baseline by ELISA technique
  percentage of A1C | 5.9 (0.5) | 5.8 (0.3) | 5.85 (0.4)
24-hours Systolic Blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3
  mmHg | 121 (8) | 119 (9) | 120 (8.5)
24-hours Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3
  mmHg | 73 (7) | 74 (7) | 73.5 (7)
Daytime Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 8 a.m. to 11 p.m. by oscillometric method Microlife WatchBP O3
  mmHg | 124 (8) | 122 (11) | 123 (9.5)
Daytime Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 8 a.m. to 11 p.m. by oscillometric method Microlife WatchBP O3
  mmHg | 75 (7) | 76 (7) | 75.5 (7)
Nightime Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 11 p.m to 8 a.m. by oscillometric method Microlife WatchBP O3
  mmHg | 114 (11) | 114 (13) | 114 (12)
Nightime Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 11 p.m to 8 a.m. by oscillometric method Microlife WatchBP O3
  mmHg | 68 (7) | 69 (8) | 68.5 (7.5)
Systolic Blood Pressure weighted Standard Deviation [Mean (Standard Deviation); unit: mmHg] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3
  mmHg | 9.2 (1.9) | 9.8 (3.3) | 9.5 (2.6)
Diastolic Blood Pressure weighted Standard Deviation [Mean (Standard Deviation); unit: mmHg] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3
  mmHg | 6.9 (1.8) | 7.7 (2.0) | 7.3 (1.9)
Coefficient of variation of 24-hours, Systolic Blood Pressure [Mean (Standard Deviation); unit: Percentage of Coefficient of variability] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3.
  Percentage of Coefficient of variability | 8.9 (2.2) | 9.2 (3.0) | 9.05 (1.91)
Coefficient of variation of 24-hours, Diastolic Blood Pressure [Mean (Standard Deviation); unit: Percentage of Coefficient of variability] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3.
  Percentage of Coefficient of variability | 11.1 (2.9) | 12.3 (2.9) | 11.7 (2.9)
Coefficient of variation of daytime, Systolic Blood Pressure [Mean (Standard Deviation); unit: Percentage of Coefficient of variability] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 8 a.m. to 11 p.m. by oscillometric method Microlife WatchBP O3
  Percentage of Coefficient of variability | 7.3 (2.2) | 8.1 (3.4) | 7.7 (2.8)
Coefficient of variation of daytime, Diastolic Blood Pressure [Mean (Standard Deviation); unit: Percentage of Coefficient of variability] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 8 a.m. to 11 p.m. by oscillometric method Microlife WatchBP O3
  Percentage of Coefficient of variability | 8.9 (2.0) | 10.0 (3.6) | 9.45 (2.8)
Coefficient of variation of nighttime, Systolic Blood Pressure [Mean (Standard Deviation); unit: Percentage of Coefficient of variability] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 11 p.m to 8 a.m. by oscillometric method Microlife WatchBP O3
  Percentage of Coefficient of variability | 8.3 (2.1) | 8.9 (3.3) | 8.6 (2.7)
Coefficient of variation of nighttime, Diastolic Blood Pressure [Mean (Standard Deviation); unit: Percentage of Coefficient of variability] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 11 p.m. to 8 a.m. by oscillometric method Microlife WatchBP O3
  Percentage of Coefficient of variability | 10.9 (4.2) | 11.9 (3.8) | 11.4 (4)
Average real variability of Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3
  mmHg | 9.5 (2.5) | 9.3 (2.0) | 9.4 (2.25)
Average real variability of Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3
  mmHg | 6.5 (1.4) | 6.6 (1.2) | 6.55 (1.3)
Number of Participants with a Nondipper circadian blood pressure pattern [Count of Participants; unit: Participants] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3
  Participants | 9 | 8 | 17
Number of Participants with a Dipper circadian blood pressure pattern [Count of Participants; unit: Participants] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3
  Participants | 5 | 4 | 9
Number of Participants with a Dipper reverse circadian blood pressure pattern [Count of Participants; unit: Participants] — Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3
  Participants | 1 | 3 | 4
Daytime Mean Arterial Pressure [Mean (Standard Deviation); unit: mmHg] — The mean arterial pressure was evaluated with ambulatory blood pressure monitoring (ABPM) from 8 a.m. to 11 p.m. by oscillometric method Microlife WatchBP O3
  mmHg | 92 (7) | 91 (8) | 91.5 (7.5)
Nighttime Mean Arterial Pressure [Mean (Standard Deviation); unit: mmHg] — The mean arterial pressure was evaluated with ambulatory blood pressure monitoring (ABPM) from 11 p.m. to 8 a.m. by oscillometric method Microlife WatchBP O3
  mmHg | 85 (8) | 84 (9) | 84.5 (8.9)
Daytime hypertensive load [Mean (Standard Deviation); unit: mmHg] — The hypertensive load was evaluated with ambulatory blood pressure monitoring (ABPM) from 8 a.m. to 11 p.m. by oscillometric method Microlife WatchBP O3
  mmHg | 30.7 (23.5) | 29.7 (29.5) | 30.2 (26.5)
Nocturnal hypertensive load [Mean (Standard Deviation); unit: mmHg] — The hypertensive load was evaluated with ambulatory blood pressure monitoring (ABPM) from 11 p.m. to 8 a.m. by oscillometric method Microlife WatchBP O3
  mmHg | 51.1 (32.3) | 45.2 (32.4) | 48.15 (32.35)

OUTCOME MEASURES:

1. Primary Outcome: 24-hours Systolic Blood Pressure at Week 12
Description: Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3
Time Frame: Week 12
Population: Each study group had 2 less participants at the end of the investigation due to withdrawal by subject, as mentioned in the participant flow, so the analysis of this outcome is calculated with those who finished the intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 117 (11) | 120 (13)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.755, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; Results showed in this section are the result of the differences between baseline and final values in dapagliflozin group; Test type: Superiority; p = 0.046, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

2. Primary Outcome: 24-hours Diastolic Blood Pressure at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 73 (8) | 75 (9)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.752, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.582, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

3. Primary Outcome: Daytime Systolic Blood Pressure at Week 12
Description: Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 8 am. to 11 p.m. by oscillometric method Microlife WatchBP O3
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 121 (11) | 122 (14)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.814, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.220, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

4. Primary Outcome: Daytime Diastolic Blood Pressure at Week 12
Description: Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 8 a.m. to p.m. by oscillometric method Microlife WatchBP O3
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 76 (9) | 77 (10)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.624, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

5. Primary Outcome: Nighttime Systolic Blood Pressure at Week 12
Description: Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 11 p.m to 8 a.m. by oscillometric method Microlife WatchBP O3
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 108 (10) | 115 (11)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.906, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.017, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

6. Primary Outcome: Nighttime Diastolic Blood Pressure at Week 12
Description: Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 11 p.m. to 8 a.m. by oscillometric method Microlife WatchBP O3
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 67 (7) | 72 (8)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.454, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.115, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

7. Primary Outcome: Systolic Blood Pressure Weighted Standard Deviation at Week 12
Description: Blood pressure variability will be evaluated with ambulatory blood pressure monitoring (ABPM) for 24 hours by oscillometric method Microlife WatchBP O3
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 9.8 (3.5) | 10.3 (2.5)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.422, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.917, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

8. Primary Outcome: Diastolic Blood Pressure Weighted Standard Deviation at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 8.0 (3.6) | 8.3 (2.0)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.650, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.108, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

9. Primary Outcome: Coefficient of Variation of 24-hours, Systolic Blood Pressure at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Coefficient of variability
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of Coefficient of variability | 9.9 (3.4) | 9.5 (1.8)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.875, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; Results showed in this section are the result of the differences between baseline and final values of waist circumference in dapagliflozin group; Test type: Superiority; p = 0.196, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

10. Primary Outcome: Coefficient of Variation of 24-hours, Diastolic Blood Pressure at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Coefficient of variability
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of Coefficient of variability | 12.3 (4.8) | 11.3 (2.2)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.552, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.087, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

11. Primary Outcome: Coefficient of Variation Daytime, Systolic Blood Pressure at Week 12
Description: Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 8 a.m to 11 p.m. by oscillometric method Microlife WatchBP O3
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Coefficient of variability
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of Coefficient of variability | 7.7 (2.4) | 8.4 (2.6)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.814, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.463, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

12. Primary Outcome: Coefficient of Variation Daytime, Diastolic Blood Pressure at Week 12
Description: Blood pressure variability was evaluated with ambulatory blood pressure monitoring (ABPM) from 8 a.m. to 11 p.m. by oscillometric method Microlife WatchBP O3
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Coefficient of variability
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of Coefficient of variability | 10.2 (4.2) | 9.2 (3.4)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.530, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.507, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

13. Primary Outcome: Coefficient of Variation Nighttime, Systolic Blood Pressure at Week 12
Description: as for outcome 6
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Coefficient of variability
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of Coefficient of variability | 8.4 (3.2) | 10.6 (4.1)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.152, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.972, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

14. Primary Outcome: Coefficient of Variation Nighttime, Diastolic Blood Pressure at Week 12
Description: as for outcome 6
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Coefficient of variability
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of Coefficient of variability | 12.3 (4.7) | 13.5 (5.0)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.152, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.158, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

15. Primary Outcome: Average Real Variability of Systolic Blood Pressure at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 10.0 (2.6) | 9.2 (2.0)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.944, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.650, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

16. Primary Outcome: Average Real Variability of Diastolic Blood Pressure at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 6.8 (1.4) | 7.0 (1.1)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.087, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.345, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

17. Primary Outcome: Number of Participants With a Nondipper Circadian Blood Pressure Pattern at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
Participants | 4 | 8
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Results showed in this section are the result of the differences between change of intervention group; Test type: Superiority; p = 0.115, Chi-squared — The threshold for statistical significance was p=0.05

18. Primary Outcome: Number of Participants With a Dipper Circadian Blood Pressure Pattern at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
Participants | 8 | 3
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Results showed in this section are the result of the differences between change of intervention groups; Test type: Superiority; p = 0.047, Chi-squared — The threshold for statistical significance was p=0.05

19. Primary Outcome: Number of Participants With a Dipper Reverse Circadian Blood Pattern at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
Participants | 1 | 2
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Results showed in this section are the result of the differences between change of intervention groups; Test type: Superiority; p = 0.539, Chi-squared — The threshold for statistical significance was p=0.05

20. Secondary Outcome: Body Weight at Week 12
Description: The body weight was measured with a bioimpedance balance
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
kg | 73 (10) | 78 (12)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.844, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.010, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

21. Secondary Outcome: Body Mass Index at Week 12
Description: Body Mas Index was calculated with the Quetelet index formula
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
kg/m^2 | 28 (2) | 29 (9)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.814, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.011, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

22. Secondary Outcome: Office Systolic Blood Pressure at Week 12
Description: Blood pressure was measured using the Omron 907-E digital sphygmomanometer (Healthcare, Inc.)
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 119 (8) | 130 (7)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.221, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

23. Secondary Outcome: Office of Diastolic Blood Pressure at Week 12
Description: Blood pressure was measured using the Omron 907-E digital sphygmomanometer (Healthcare, Inc.)
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 75 (6) | 82 (8)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.461, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.011, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

24. Secondary Outcome: Fasting Plasma Glucose Levels at Week 12
Description: The fasting glucose levels was evaluated with enzymatic/colorimetric techniques
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 5.8 (0.5) | 6.1 (0.7)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.285, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

25. Secondary Outcome: 2-hours Plasma Glucose After a Oral Glucose Tolerance Test at Week 12
Description: 2-hours plasma glucose after a oral glucose tolerance test (75 g of glucose load). Glucose was evaluated with enzymatic/ colorimetric technique
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 7.8 (1.8) | 8.3 (2.8)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.701, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.081, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

26. Secondary Outcome: Glycated Hemoglobin A1c (A1C) at Week 12
Description: A1C was evaluated by Enzyme-Linked ImmunoSorbent Assay (ELISA)
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of A1C
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
percentage of A1C | 5.4 (0.4) | 5.9 (0.4)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.581, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; Results showed in this section are the result of the differences between baseline and final values of HDL-cholesterol on dapagliflozin group; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

27. Secondary Outcome: Daytime Mean Arterial Pressure at Week 12
Description: The mean arterial pressure was evaluated with ambulatory blood pressure monitoring (ABPM) from 8 a.m. to 11 p.m. by oscillometric method Microlife WatchBP O3
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 92 (11) | 92 (10)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.727, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.451, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

28. Secondary Outcome: Nighttime Mean Arterial Pressure at Week 12
Description: The Mean Arterial Pressure was evaluated with ambulatory blood pressure monitoring (ABPM) from 11 p.m. to 8 a.m. by oscillometric method Microlife WatchBP O3
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 84 (9) | 87 (9)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.463, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.043, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

29. Secondary Outcome: Daytime Hypertensive Load at Week 12
Description: The hypertensive load was evaluated with ambulatory blood pressure monitoring (ABPM) from 8 a.m. to 11 p.m. by oscillometric method Microlife WatchBP O3
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of hypertensive load
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
percentage of hypertensive load | 28.6 (29.8) | 34.1 (35.7)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.807, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.754, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

30. Secondary Outcome: Nocturnal Hypertensive Load at Week 12
Description: The Hypertensive Load was evaluated with ambulatory blood pressure monitoring (ABPM) from 11 p.m. to a.m. by oscillometric method Microlife WatchBP O3
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of hypertensive load
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
percentage of hypertensive load | 38.1 (32.0) | 52.0 (32.0)
Statistical Analysis 1: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values in placebo group; Test type: Superiority; p = 0.507, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Dapagliflozin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.015, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

31. Secondary Outcome: Number of Participants With Prediabetes at Week 12
Description: Prediabetes was diagnosed with the criteria of the American Diabetes Association.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
Participants | 7 | 2
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Results showed in this section are the result of the differences between intervention groups; Test type: Superiority; p = 0.039, Fisher Exact — The threshold for statistical significance was p=0.05

32. Secondary Outcome: Number of Participants With Prehypertension at Week 12
Description: Prehypertension was diagnosed with the criteria of the Eighth Joint National Committee.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
Participants | 7 | 1
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Results showed in this section are the result of the differences between intervention groups; Test type: Superiority; p = 0.011, Fisher Exact

33. Secondary Outcome: Number of Participants With Prediabetes Plus Prehypertension at Week 12
Description: Criteria of the American Diabetes Association and Eighth Joint National Committee were used to diagnosed prediabetes and prehypertension.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 13 | 13
Participants | 4 | 0
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Results showed in this section are the result of the differences between intervention groups; Test type: Superiority; p = 0.096, Fisher Exact — The threshold for statistical significance was p=0.05

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 12 weeks
Arm/Group | Dapagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=15) | Placebo (N=15)
Cervicovaginal infection (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infections (Renal and urinary disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT03006471/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT03006471/Prot_SAP_001.pdf